CLINICAL TRIAL: NCT03506932
Title: A Randomized, Controlled, Cross-over Trial Examining the Effect of Yellow Pea Flour in Bread on Post-prandial Glycaemic Response in Healthy Adults
Brief Title: Effect of Pea Flour in Bread on Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government); University of Manitoba (Other); Saskatchewan Pulse Growers (Other)
Responsible Party: Principal Investigator, Dr. Heather Blewett, Principal Investigator, St. Boniface Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HS21603 (B2018:026); RRC/2018/1748 (Other: St. Boniface Hopsital Research Review Committee)
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Post-prandial Glycaemic Response
Keywords: blood sugar; insulin; peas; bread; metabolites
MeSH Terms: conditions — Insulin Resistance | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Untreated (Experimental): Bread containing 20% yellow pea flour.
  Interventions: Dietary Supplement: Untreated
- Heat treated with 0% moisture (Experimental): Bread containing 20% yellow pea flour.
  Interventions: Dietary Supplement: Heat treated with 0% moisture
- Heat treated with 10% moisture (Experimental): Bread containing 20% yellow pea flour.
  Interventions: Dietary Supplement: Heat treated with 10% moisture
- Wheat (Active Comparator): Bread made with 100% wheat flour
  Interventions: Dietary Supplement: Wheat

INTERVENTIONS:
Dietary Supplement: Untreated — Bread made with 20% yellow pea flour that was untreated.
  Arms: Untreated
Dietary Supplement: Heat treated with 0% moisture — Bread made with 20% yellow pea flour that was heat treated with 0% moisture.
  Arms: Heat treated with 0% moisture
Dietary Supplement: Heat treated with 10% moisture — Bread made with 20% yellow pea flour that was heat treated with 10% moisture.
  Arms: Heat treated with 10% moisture
Dietary Supplement: Wheat — Bread made with 100% wheat
  Arms: Wheat

SUMMARY:
This study's overall goal is to investigate methods to improve the acceptability of pulse containing foods that provide a health benefit to consumers. The health benefits we are testing are post-prandial blood glucose attenuation and appetite related sensations in healthy human volunteers.

DETAILED DESCRIPTION:
A randomized, controlled, cross-over study designed to examine the post-prandial glycaemic response, metabolism of bioactives and appetite related sensations to 20% incorporation of yellow pea flour (untreated, heat treated with 0% moisture and heat treated with 10% moisture) into bread will be conducted at the I.H. Asper Clinical Research Institute in Winnipeg, Manitoba. Eligible participants who have provided consent will be asked to attend 4 clinic visits in a fasted state. Participants will be given bread containing 20% yellow pea flour at 3 visits and bread with 100% wheat flour at 1 visit. At each visit participants will provide 7 venous blood samples via indwelling catheter, 7 capillary blood samples via finger poke, 2 urine samples, 5 questionnaires about their appetite and a questionnaire about the acceptability of the products. Each visit will last approximately 3h and be separated by 3-14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy male or female, between the age of 18-40 years;
2. Body mass index (BMI) 18.5-30.0 kg/m2;
3. Habitually consume breakfast, lunch and dinner in the morning, mid-day and evening, respectively;
4. Willing to provide informed consent;
5. Willing/able to comply with the requirements of the study.

Exclusion Criteria:

1. Pregnant or lactating;
2. Medical history of diabetes mellitus, fasting blood glucose ≥6.1 mmol/L, HbA1c ≥6.0%, or use of insulin or oral medication to control blood sugar;
3. Medical history of cardiovascular disease;
4. Systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg;
5. Fasting plasma total cholesterol >7.8 mmol/L;
6. Fasting plasma HDL <0.9 mmol/L;
7. Fasting plasma LDL >5.0 mmol/L;
8. Fasting plasma triglycerides >2.3 mmol/L;
9. Major surgery within the last 3 months;
10. Medical history of inflammatory disease (ie. Systemic lupus erythematosis, rheumatoid arthritis, psoriasis) or use of any corticosteroid medications within 3 months;
11. Medical history of liver disease or liver dysfunction (defined as plasma aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥3 times the upper limit of normal (ULN));
12. Medical history of kidney disease or kidney dysfunction (defined as blood urea nitrogen and creatinine ≥3 times the ULN));
13. Presence of a gastrointestinal disorder, daily use of any stomach acid-lowering medications or laxatives (including fibre supplements) within the past month or antibiotic use within the past 6 weeks;
14. Active treatment for any type of cancer within 1 year prior to study start;
15. Shift worker (a system of employment where an individual's normal hours of work are in part, outside the period of normal working day; 6am and 8pm);
16. Smoking, use of tobacco or a nicotine replacement product, and cannabis in any form (within the last 3 months);
17. Allergies to peas or wheat;
18. Aversion or unwillingness to eat study foods;
19. Consuming >4 servings of pulses per week;
20. Use of any prescription or non-prescription drug, herbal or nutritional supplement known to affect glycaemia or appetite;
21. Participation in another clinical trial, current or in the past 4 weeks;
22. Unstable body weight (defined as >5% change in 3 months) or actively participating in a weight loss program.
23. Other medical, psychiatric, or behavioral factors that in the judgment of the principal Investigator may interfere with study participation or the ability to follow the intervention protocol;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Post-prandial glucose | 120 minutes
  incremental area under the curve (iAUC) for glucose
Post-prandial insulin | 120 minutes
  iAUC insulin

SECONDARY OUTCOMES:
Urinary metabolite profile | 120 minutes
  Concentration of metabolites in urine
Plasma metabolite profile | 120 minutes
  Concentration of metabolites in plasma

OTHER OUTCOMES:
Hunger | 120 minutes
  Area under the curve (AUC) using visual analog scales
Fullness | 120 minutes
  AUC using visual analog scales
Desire to eat | 120 minutes
  AUC using visual analog scales
Prospective consumption | 120 minutes
  AUC using visual analog scales
Acceptability of test products | 15 minutes
  Ratings of color, aroma, flavor, texture and frequency of eating
Gastrointestinal effects | 24 hours
  Incidence of gastrointestinal side effects

CONTACTS AND LOCATIONS:
Overall Officials: Heather Blewett, PhD, Principal Investigator — Agriculture and Agri-Food Canada
Locations (1):
- I. H. Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the time the data is collected until manuscript is accepted for publication.
Access Criteria: Michel Aliani and Sora Ludwig will have access to data necessary for manuscript preparation.

REFERENCES:
- [Background] Sievenpiper JL, Kendall CW, Esfahani A, Wong JM, Carleton AJ, Jiang HY, Bazinet RP, Vidgen E, Jenkins DJ. Effect of non-oil-seed pulses on glycaemic control: a systematic review and meta-analysis of randomised controlled experimental trials in people with and without diabetes. Diabetologia. 2009 Aug;52(8):1479-95. doi: 10.1007/s00125-009-1395-7. Epub 2009 Jun 13. PMID 19526214
- [Background] Marinangeli CP, Jones PJ. Chronic intake of fractionated yellow pea flour reduces postprandial energy expenditure and carbohydrate oxidation. J Med Food. 2011 Dec;14(12):1654-62. doi: 10.1089/jmf.2010.0255. PMID 22145774
- [Background] Robinson DS, Wu Z, Domoney C, Casey R. Lipoxygenases and the quality of foods. Food Chem 54:33-43,1995.
- [Background] Rackis JJ, Sessa DJ, Honig DH. Flavor problems of vegetable food proteins. J Am Oil Chem Soc 56(3):262-71,1979.
- [Background] Shariati-Ievari S, Ryland D, Edel A, Nicholson T, Suh M, Aliani M. Sensory and Physicochemical Studies of Thermally Micronized Chickpea (Cicer arietinum) and Green Lentil (Lens culinaris) Flours as Binders in Low-Fat Beef Burgers. J Food Sci. 2016 May;81(5):S1230-42. doi: 10.1111/1750-3841.13273. Epub 2016 Mar 15. PMID 26990186
- [Background] Mitzak, M. 2007. Method for heat treatment of powdery materials (Google Patents).
- [Background] Jenkins DJ, Thorne MJ, Camelon K, Jenkins A, Rao AV, Taylor RH, Thompson LU, Kalmusky J, Reichert R, Francis T. Effect of processing on digestibility and the blood glucose response: a study of lentils. Am J Clin Nutr. 1982 Dec;36(6):1093-101. doi: 10.1093/ajcn/36.6.1093. PMID 6293296
- [Background] Li H, Song F, Xing J, Tsao R, Liu Z, Liu S. Screening and structural characterization of alpha-glucosidase inhibitors from hawthorn leaf flavonoids extract by ultrafiltration LC-DAD-MS(n) and SORI-CID FTICR MS. J Am Soc Mass Spectrom. 2009 Aug;20(8):1496-503. doi: 10.1016/j.jasms.2009.04.003. Epub 2009 Apr 14. PMID 19443236
- [Background] Habtemariam S. A-glucosidase inhibitory activity of kaempferol-3-O-rutinoside. Nat Prod Commun. 2011 Feb;6(2):201-3. PMID 21425674
- [Background] Blundell J, de Graaf C, Hulshof T, Jebb S, Livingstone B, Lluch A, Mela D, Salah S, Schuring E, van der Knaap H, Westerterp M. Appetite control: methodological aspects of the evaluation of foods. Obes Rev. 2010 Mar;11(3):251-70. doi: 10.1111/j.1467-789X.2010.00714.x. Epub 2010 Jan 29. PMID 20122136
- [Background] European Food Safety Authority. Guidance on the scientific requirements for health claims related to appetite ratings, weight management, and blood glucose concentrations. EFSA Journal. 10(3):2604, 2012.
- [Background] Health Canada. Draft guidance document: Satiety health claims on food [Internet].; 2012. Available from: http://www.hc-sc.gc.ca/fn-an/consult/satiety-satiete/document-consultation-eng.php
- [Background] Ames N, Blewett H, Storsley J, Thandapilly SJ, Zahradka P, Taylor C. A double-blind randomised controlled trial testing the effect of a barley product containing varying amounts and types of fibre on the postprandial glucose response of healthy volunteers. Br J Nutr. 2015 May 14;113(9):1373-83. doi: 10.1017/S0007114515000367. Epub 2015 Apr 8. PMID 25850814
- [Background] Brouns F, Bjorck I, Frayn KN, Gibbs AL, Lang V, Slama G, Wolever TM. Glycaemic index methodology. Nutr Res Rev. 2005 Jun;18(1):145-71. doi: 10.1079/NRR2005100. PMID 19079901
- [Background] Rabiee A, Magruder JT, Grant C, Salas-Carrillo R, Gillette A, DuBois J, Shannon RP, Andersen DK, Elahi D. Accuracy and reliability of the Nova StatStrip(R) glucose meter for real-time blood glucose determinations during glucose clamp studies. J Diabetes Sci Technol. 2010 Sep 1;4(5):1195-201. doi: 10.1177/193229681000400519. PMID 20920440
- [Background] Public Health Agency of Canada and the Canadian Institute for Health Information. Obesity in Canada: A joint report from the Public Health Agency of Canada and the Canadian institute for health information. Government of Canada; 2011.
- [Background] Public Health Authority of Canada. Diabetes in Canada: Facts and figures from a public health perspective. 2011.